CLINICAL TRIAL: NCT00678080
Title: A Randomized, Controlled Trial of Metformin Versus Insulin in Women With Type 2 Diabetes Mellitus During Pregnancy in a Population With Severe Health Disparities
Brief Title: Metformin Versus Insulin in Pregnant Women With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jerrie Refuerzo, Associate Professor - Ob/Gyn Maternal Fetal, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-08-0015
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy Complications
Keywords: Type 2 diabetes mellitus; Pregnancy; Metformin; Insulin; Pregnant women
MeSH Terms: conditions — Pregnancy Complications; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin therapy as prescribed by their health care provider
  Interventions: Drug: Metformin
- Insulin (Active Comparator): Insulin as prescribed by their health care provider
  Interventions: Drug: Insulin (NPH and Regular)

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg orally daily increased as needed to maintain glycemic control until a maximum of 2500 daily
  Other Names: Glucophage
  Arms: Metformin
Drug: Insulin (NPH and Regular) — Insulin will be administered based on maternal gestational age and maternal weight using NPH and Regular insulin. It will be administered subcutaneously 3 times a day
  Arms: Insulin

SUMMARY:
Pregnant women with type 2 diabetes mellitus (T2DM) are at increased risk for miscarriages, birth defects, large infants, and stillbirths. Maintaining blood sugars in the normal range decreases these pregnancy complications. We hypothesize that metformin will achieve similar levels of blood sugar control compared to insulin. In doing so, metformin will prevent the increased risk of pregnancy complications associated with T2DM in pregnancy. We propose a pilot study of a randomized, controlled trial of metformin versus insulin in the treatment of T2DM during pregnancy.

DETAILED DESCRIPTION:
Pregnant women with type 2 diabetes mellitus (T2DM) are at increased risk for miscarriages, birth defects, large infants, and stillbirths. Maintaining blood sugars in the normal range decreases these pregnancy complications. Currently, insulin is the primary medication used to treat pregnant women with T2DM. However, it is administered by injection several times a day and compliance is low in health disparity populations with high rates of obesity and diabetes. Insulin also has the potential to lead to dangerously low blood sugars. Metformin is a medication than can be administered as pills and is not associated with dangerous low blood sugars. In addition, this insulin sensitizer is the medication of choice for women who are obese and have T2DM outside of pregnancy. We hypothesize that metformin will achieve similar levels of blood sugar control compared to insulin. In doing so, metformin will prevent the increased risk of pregnancy complications associated with T2DM in pregnancy. The aims of this study is to determine if in pregnant women with T2DM, metformin achieves similar glycemic control, and similar maternal and neonatal outcomes when compared to insulin. We propose a pilot study of a randomized, controlled trial of metformin versus insulin in the treatment of T2DM during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* The onset of T2DM for less than 10 years prior to the onset of pregnancy by patient history
* Treatment with diet or oral hypoglycemic agents prior to pregnancy.
* Pregnancies less than 20 weeks of pregnancy. This gestational age was chosen to include those women who initiated prenatal care in the second trimester, but still have the ability to improve their hemoglobin A1C (primary outcome) with medical therapy prior to delivery.
* Newly diagnosed diabetes in the first 20 weeks of pregnancy. These women likely have had diabetes prior to the onset of pregnancy. They do not qualify for the diagnosis of gestational diabetes which is typically made after 20 weeks of pregnancy. Diagnosis will be made based on an elevated fasting blood glucose greater than 105 mg/dL, a 50 gram glucola result greater than 200 mg/dL or an abnormal 3 hour glucola test prior to 20 weeks of pregnancy. An abnormal 3-hour glucola test is defined as 2 out of 4 abnormal values.
* Hemoglobin A1C <9%

Exclusion Criteria:

* Gestational age greater than 20 weeks
* Multiple gestations (twins or more gestations)
* Type 1 diabetes by patient history
* Known fetal chromosomal or structural defects
* Contraindications to the use of metformin including renal disease, liver disease, prior myocardial infarction or sepsis.
* Those with a hemoglobin A1C greater than 9%.
* On insulin at the start of pregnancy

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrie S Refuerzo, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - Valley Baptist Hospital, Brownsville, Texas
  - Lyndon B Johnson Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin therapy
  Metformin: Metformin 500 mg orally daily increased as needed to maintain glycemic control until a maximum of 2500 daily
- Insulin: Insulin
  Insulin (NPH and Regular): Insulin will be administered based on maternal gestational age and maternal weight using NPH and Regular insulin. It will be administered subcutaneously 3 times a day
Period: Overall Study
Arm/Group | Metformin | Insulin
Started | 11 | 14
Completed | 8 | 13
Not Completed | 3 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Insulin | Total
Number analyzed (Participants) | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (5.5) | 32.3 (4.3) | 31.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 6 | 10
  African American | 3 | 4 | 7
  Hispanic | 0 | 1 | 1
  Other | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Achieved a Hemoglobin A1C <7%
Description: The hemoglobin A1c level is an indicator of glycemic control-it indicates the average level of blood sugar over the past 2 to 3 months. Hemoglobin A1c levels 6.5% and higher indicate diabetes.
Time Frame: during third trimester
Population: During the third trimester, hemoglobin A1c levels were obtained for only 5 in the metformin arm and 12 in the insulin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 5 | 12
Participants | 5 | 12

2. Secondary Outcome: Body Mass Index
Time Frame: at the time of delivery
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
kg/m^2 | 35.9 (5.2) | 40.1 (8.4)

3. Secondary Outcome: Number of Participants With Hypoglycemia
Description: Defined as hypoglycemia as documented by neonatal chart based on health care provider description
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Who Failed Metformin Therapy
Description: Those whose glucose levels were above target range thereby needing insulin therapy
Time Frame: Duration of pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 0
Participants | 0 |

5. Secondary Outcome: Number of Participants Who Had a Cesarean Section
Time Frame: At the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
Participants | 4 | 6

6. Secondary Outcome: Number of Participants With Fetus With Macrosomia
Time Frame: At the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
Participants | 0 | 1

7. Secondary Outcome: Number of Participants With Shoulder Dystocia
Time Frame: At the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
Participants | 1 | 0

8. Secondary Outcome: Number of Participants Who Had a Newborn With Respiratory Distress Syndrome
Time Frame: Neonatal period
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
Participants | 1 | 3

9. Secondary Outcome: Number of Participants With Newborns Who Needed Neonatal Dextrose
Time Frame: Neonatal period
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 8 | 13
Participants | 0 | 1

10. Primary Outcome: The Number of Participants Who Achieved a Hemoglobin A1C <7%
Description: as for outcome 1
Time Frame: at the time of delivery
Population: At the time of delivery, hemoglobin A1c levels were obtained for only 5 in the metformin arm and 8 in the insulin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 5 | 8
Participants | 5 | 7

ADVERSE EVENTS:
Arm/Group | Metformin | Insulin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 0/8 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No